CLINICAL TRIAL: NCT01059318
Title: An Exploratory, Open-label, Non-randomized, Within-patient Multiple Dose-escalation Safety, Tolerability, PK and Efficacy Trial of RAD001 (Everolimus) in Patients With Lymphangioleiomyomatosis
Brief Title: A Study to Determine the Safety and Effectiveness of RAD001 (Everolimus) in Patients With Lymphangioleiomyomatosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001X2201; 2010-019825-32 (EudraCT Number)
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Lymphangioleiomyomatosis
Keywords: Lymphangioleiomyomatosis,; High Resolution CT scan,; chest x-ray,; 6 minute walk test,; pulse oximetry,; renal MRI,; Pikometer
MeSH Terms: conditions — Lymphangioleiomyomatosis | interventions — Everolimus

ARMS (1):
- Everolimus (Experimental): All patients received a starting dose of everolimus 2.5mg/day for 4 weeks, followed by a dose of 5 mg/day for 4 weeks and finally a dose of 10mg/day for 18 weeks.
  The 26 week treatment period was followed by an optional extension period wherein patients continued therapy until the last patient had completed 26-weeks of treatment. The longest period a patient participated in the study was 62 weeks.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Everolimus was formulated as tablets in strengths of 2.5mg, 5mg and 10mg.
  Other Names: RAD001

SUMMARY:
This was an exploratory study to determine whether escalating doses of RAD001 (everolimus) were safe and effective in patients with Lymphangioleiomyomatosis

DETAILED DESCRIPTION:
In addition to the data collected in this study, historical data from 43 patients treated with placebo from the multicenter trial of sirolimus in LAM (MILES) study (NCT00414648) were down weighted to an effective sample size of 18 for comparison of FEV1 and FVC endpoints. Reference to the publication of the MILES study has been provided under "Result Publication".

ELIGIBILITY:
Inclusion Criteria:

* Female aged >/= 18 years with a diagnosis of LAM
* Pulmonary function abnormalities as follows:
* FEV1 of ≤ 80% of the predicted value following administration of a standard dose of a short acting β2-agonist (*200 µg Salbutamol, measured between 10 and 15 minutes of inhalation) OR
* FEV1 < 90% of the predicted value of bronchodilator following administration of a standard dose of a short acting β2-agonist (*200 µg Salbutamol, measured between 10 and 15 minutes of inhalation) and DLco (uncorrected) <80% predicted.
* Female patients including those of childbearing potential will be included in this study.
* Negative pregnancy test at screening and baseline

Exclusion Criteria:

* FEV1<50% of predicted post-bronchodilator.
* Change in FVC (ml) > ± 15% of screening value at baseline visit (not less than 14d after screening visit).
* Use of any medicine containing estrogen in the 4 months prior to the screening visit and for the duration of the study
* Significant hematologic, renal, hepatic laboratory abnormality or amylase > 1.5x the upper limit of the normal range at the screening or baseline visits
* Fasting blood glucose > 126mg/dl or random blood glucose >200mg/dl at screening and/or baseline
* Recent surgery (involving entry into a body cavity or requiring sutures) within 2 months of the screening visit or any evidence of unhealed surgical wound.
* Uncontrolled hyperlipidemia (defined as persistent elevation of total cholesterol or triglycerides >6.5nM/L) or a history of clinical atherosclerotic disease including heart attack, angina, peripheral vascular disease or stroke.
* Previous organ transplantation
* Inability to give informed consent
* Inability to perform pulmonary function or 6 minute walk tests and imaging assessments

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (2):
  - Center for LAM Research and Clinical Care, Boston, Massachusetts
  - University of Cincinnati, Department of Internal Medicine, Pulmonary, Critical Care & Sleep Medicine,, Cincinnati, Ohio
- Novartis Investigative Site, Lyon, France
- Novartis Investigative Site, Milan, Italy

REFERENCES:
- [Result] McCormack FX, Inoue Y, Moss J, Singer LG, Strange C, Nakata K, Barker AF, Chapman JT, Brantly ML, Stocks JM, Brown KK, Lynch JP 3rd, Goldberg HJ, Young LR, Kinder BW, Downey GP, Sullivan EJ, Colby TV, McKay RT, Cohen MM, Korbee L, Taveira-DaSilva AM, Lee HS, Krischer JP, Trapnell BC; National Institutes of Health Rare Lung Diseases Consortium; MILES Trial Group. Efficacy and safety of sirolimus in lymphangioleiomyomatosis. N Engl J Med. 2011 Apr 28;364(17):1595-606. doi: 10.1056/NEJMoa1100391. Epub 2011 Mar 16. PMID 21410393
- [Derived] Goldberg HJ, Harari S, Cottin V, Rosas IO, Peters E, Biswal S, Cheng Y, Khindri S, Kovarik JM, Ma S, McCormack FX, Henske EP. Everolimus for the treatment of lymphangioleiomyomatosis: a phase II study. Eur Respir J. 2015 Sep;46(3):783-94. doi: 10.1183/09031936.00210714. Epub 2015 Jun 25. PMID 26113676

RESULTS

PARTICIPANT FLOW:
Groups:
- Everolimus: All patients received a starting dose of everolimus 2.5mg/day for 4 weeks, followed by a dose of 5 mg/day for 4 weeks and finally a dose of 10mg/day for 18 weeks. The 26 week treatment period was followed by an optional extension period wherein patients continued therapy until the last patient had completed 26-weeks of treatment. The longest period a patient participated in the study was 62 weeks.
  Everolimus : Everolimus was formulated as tablets in strengths of 2.5mg, 5mg and 10mg.
Period: Core Study (26 Week)
Arm/Group | Everolimus
Started | 24 (This is safety set and Pharmacodynamic set)
Everolimus 2.5 mg for 4 Weeks | 24
Everolimus 5 mg for 4 Weeks | 24
Everolimus 10 mg for 18 Weeks | 24
Pharmacokinetics (PK) Analysis Set | 16 (For 8 patients plasma rather than whole blood sample was collected, hence excluded from PK set.)
Completed | 20
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Period: Extension (36 Week)
Arm/Group | Everolimus
Started | 20
Completed | 17
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: Everolimus arm has all patients who received study drug that is the safety analysis set.
Arm/Group | Everolimus
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Vascular Endothelial Growth Factor-D (VEGF-D) Concentrations
Description: Blood samples (1 mL) for determination of VEGF-D were collected from a forearm vein (direct venipuncture or from an indwelling cannula) and 2 aliquots of serum were collected. VEGF-D levels were determined from only 1 of the 2 serum aliquots, with the second acting as a back-up. A serum VEGF-D >800 pg/mL level supports a diagnosis of Lymphangioleiomyomatosis (LAM)
Time Frame: Baseline, 26 weeks
Population: Pharmacodynamic analysis included patients who received study drug without any major protocol violation. Same patients in different dose groups were included in this analysis with available data.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Everolimus 2.5 mg/Day: All patients received a starting dose of everolimus 2.5mg/day for first 4 weeks.
- Everolimus 5 mg/Day: Patients from 2.5 mg/day up-titrated after 4 weeks and followed by a dose of 5 mg/day for another 4 weeks.
- Everolimus 10 mg/Day: Patients who had received 2.5 mg/day for first 4 weeks, up titrated to 5 mg/day and continued for another 4 weeks, again up-titrated to 10 mg/day for 18 weeks.
Arm/Group | Everolimus 2.5 mg/Day | Everolimus 5 mg/Day | Everolimus 10 mg/Day
Number analyzed (Participants) | 21 | 22 | 22
pg/mL | -464.3 (745.23) | -1113.2 (1468.9) | -1771.7 (2091.6)

2. Primary Outcome: Mean Trough (C0,ss) and Peak (C2,ss) Drug Concentration at Steady State
Description: Venous blood samples (2 mL) for pharmacokinetic evaluation were collected pre dose and 2 hours post dose at preselected visits.
Time Frame: pre-dose and at 2 hour post dose at week 26
Population: Pharmacokinetics analysis set. Patients with measurable data at particular time points were included in this analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Everolimus 2.5 mg/Day | Everolimus 5 mg/Day | Everolimus 10 mg/Day
Number analyzed (Participants) | 16 | 16 | 16
ng/mL
  Trough (C0, ss): number analyzed (Participants) | 13 | 14 | 11
  Trough (C0, ss) | 3.1 (1.33) | 5.8 (3.02) | 11.0 (3.45)
  Peak (C2, ss): number analyzed (Participants) | 13 | 16 | 10
  Peak (C2, ss) | 12.1 (3.56) | 22.6 (7.22) | 45.7 (12.52)

3. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC)
Description: All spirometry evaluation followed recommendations of the Standardization of Lung Function Testing. All spirometry maneuvers were performed in sitting position whilst wearing nose clips. At least three acceptable maneuvers were performed for each time point, and results met within-test and between-test criteria for acceptability. The highest value was obtained of FVC from any of the three maneuvers that met acceptability criteria. Change from baseline in FVC was compared between everolimus and historical placebo data from multicenter trial of sirolimus in LAM. (MILES NCT00414648) due to absence of placebo group in this current study on a rare lung disease. These two studies had different study designs, so the change from baseline to 6 months (26 weeks) in MILES study was estimated from the publicly reported rate of change per month to provide a meaningful comparison. This historical control be can be viewed on the Novartis Clinical Trial Results website.
Time Frame: Baseline, 26 weeks
Population: Pharmacodynamic analysis set for everolimus reporting arm. Patients with both baseline and 26 weeks assessment were included in this analysis.
Measure: Mean (95% Confidence Interval); unit: mL
Groups:
- Everolimus: All patients received a starting dose of everolimus 2.5mg/day for 4 weeks, followed by a dose of 5 mg/day for 4 weeks and finally a dose of 10mg/day for 18 weeks.
  Everolimus : Everolimus was formulated as tablets in strengths of 2.5mg, 5mg and 10mg.
Arm/Group | Everolimus
Number analyzed (Participants) | 23
mL | 10 [-111 to 132]
Statistical Analysis 1: Comparison: Everolimus; Proof of Concept was proposed as follows: * 90% level of proof that difference in FVC change from baseline everolimus vs. Historical Placebo Control arm from MILES study > 0 mL * 50% level of proof that difference in FVC change from baseline everolimus vs. Historical Placebo Control arm from MILES study >= 100 mL Historical data from 43 patients treated with placebo from the MILES study were down weighted to an effective sample size of 18 for comparison; Test type: Superiority or Other; Bayesian analysis; A Bayesian posterior distribution of the treatment effect at 26 weeks was evaluated using a non-informative prior; Mean Difference (Final Values) = 76, 95% CI 2-sided [-45 to 196] — MILES study and current study had different study designs, so change from baseline to 26 weeks in MILES study was estimated from the publicly reported rate of change per month in order to provide a meaningful comparison based on Bayesian analysis

4. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1)
Description: All spirometry evaluation followed the recommendations of the Standardization of Lung Function Testing. All spirometry maneuvers were performed in the sitting position whilst wearing nose clips. At least three acceptable maneuvers were performed for each time point, and the results met within-test and between-test criteria for acceptability. The highest value was obtained of FEV1 from any of the three maneuvers that met acceptability criteria.
  Change from baseline in FEV1 was compared between everolimus and historical placebo data from the MILES study (NCT00414648) due to the absence of a placebo group in this current study on a rare lung disease. These two studies had different study designs, so the change from baseline to 6 months (26 weeks) in MILES study was estimated from the publicly reported rate of change per month in order to provide a meaningful comparison. This historical control can be viewed on the Novartis Clinical Trial Results website.
Time Frame: Baseline, 26 weeks
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Everolimus
Number analyzed (Participants) | 23
mL | 114 [11 to 217]
Statistical Analysis 1: Comparison: Everolimus; Proof of Concept was proposed as follows: * 90% level of proof that difference in FEV1 change from baseline everolimus vs. Historical Placebo Control arm from MILES study > 0 mL * 50% level of proof that difference in FEV1 change from baseline everolimus vs. Historical Placebo Control arm from MILES study >= 100 mL Historical data from 43 patients treated with placebo from the MILES study were down weighted to an effective sample size of 18 for comparison; Test type: Superiority or Other; Bayesian analysis; A Bayesian posterior distribution of the treatment effect at 26 weeks was evaluated using a non-informative prior; Mean Difference (Final Values) = 186, 95% CI 2-sided [93 to 279] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Change From Baseline in Extended Pulmonary Function Testing
Description: Extended pulmonary function testing such as Total Lung Capacity (TLC), Thoracic Gas Volume (TGV), Residual Volume (RV) were measured using a body plethysmograph
Time Frame: Baseline, 26 weeks
Population: Pharmacodynamic analysis set. Patients with both baseline and 26 weeks assessment were included in the analysis.
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Everolimus
Number analyzed (Participants) | 22
Liters (L)
  TLC | 0.199 (0.8645)
  TGV | 0.267 (1.0368)
  RV | 0.169 (0.9055)

6. Secondary Outcome: Change From Baseline in Carbon Monoxide Diffusing Capacity (DLCO)
Description: Carbon Monoxide Diffusing Capacity (DLCO) one of the extended pulmonary function testing which was also measured using a body plethysmograph.
Time Frame: Baseline, 26 weeks
Population: Pharmacodynamic analysis set. Patients with both baseline and 26 weeks assessment were included in the analysis.
Measure: Mean (Standard Deviation); unit: ml/min/mmHg
Arm/Group | Everolimus
Number analyzed (Participants) | 22
ml/min/mmHg | -0.782 (1.5351)

7. Secondary Outcome: Change From Baseline in 6-minute Walk Test Score to Measure Exercise Capacity
Description: A standardized 6-minute walk test (6MWT) was performed in accordance with the guidelines of the American Thoracic Society 2002. The test was done about the same time of day to avoid diurnal variation in an environment that had an adequate temperature to avoid additional burden to the patient due to heat or cold air. The distance walked in six minutes (6MWD) was recorded.
Time Frame: Baseline, 26 weeks
Population: Pharmacodynamic analysis set. Patients with both baseline and 26 weeks assessment were included in the analysis.
Measure: Mean (Standard Deviation); unit: meters (m)
Arm/Group | Everolimus
Number analyzed (Participants) | 23
meters (m) | 46.9 (115.30)

8. Secondary Outcome: Change From Baseline in Oxygen Saturation
Description: Oxygen saturation means the amount of oxygen in blood stream. Oxygen saturation was measured by using a Pulse Oximeter.
Time Frame: Baseline, 26 weeks
Population: Pharmacodynamic analysis set. Patients with both baseline and 26 weeks assessment were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of oxygen
Arm/Group | Everolimus
Number analyzed (Participants) | 23
percentage of oxygen | 0.8 (2.13)

ADVERSE EVENTS:
Description: Safety set includes all the patients who had received at least one dose of study drug.
Arm/Group | Everolimus
Serious Adverse Events (participants affected / at risk) | 8/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=24)
Cardiac failure (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Pneumocystis jiroveci infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=24)
Abdominal pain upper (Gastrointestinal disorders) | 2
Aphthous stomatitis (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 7
Haemorrhoids (Gastrointestinal disorders) | 3
Mouth ulceration (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 7
Stomatitis (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 7
Non-cardiac chest pain (General disorders) | 5
Oedema peripheral (General disorders) | 6
Pyrexia (General disorders) | 2
Bronchitis (Infections and infestations) | 2
Ear infection (Infections and infestations) | 2
Furuncle (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 4
Oral herpes (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 2
Vulvovaginal mycotic infection (Infections and infestations) | 2
Post-traumatic pain (Injury, poisoning and procedural complications) | 2
Gamma-glutamyltransferase increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 9
Insomnia (Psychiatric disorders) | 3
Dysmenorrhoea (Reproductive system and breast disorders) | 2
Menorrhagia (Reproductive system and breast disorders) | 2
Menometorrhagia (Reproductive system and breast disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.